CLINICAL TRIAL: NCT05486078
Title: Evaluation of the Efficacy of the Use of a Type I Collagen-based MD Tissue Collagen Medical Device in the Infiltrative Treatment of Greater Trochanter Pain Syndrome (GTPS) "MEDANTRO PILOT STUDY"
Brief Title: Evaluation of the Efficacy of the Use MD Tissue Collagen Medical Device in the Infiltrative Treatment of Greater Trochanter Pain Syndrome (GTPS)
Acronym: MEDANTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guna S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDG2020711
Record Dates: First submitted 2022-07-04; First posted 2022-08-03 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Greater Trochanteric Pain Syndrome; GTPS - Greater Trochanteric Pain Syndrome; Tendon Disorder; Pertrochanteric Fracture; Gluteal Tendinitis; Gluteal Muscles
Keywords: MD-Tissue Collagen Medical; Ecoguide; Biomechanical; Modified Harris Hip Score; Numeric Rating Scale; Type I collagen
MeSH Terms: conditions — Tendinopathy; Osteogenesis Imperfecta, Type IV

STUDY DESIGN:
Intervention Model Description: One sample study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD-Tissue Medical Device (Experimental)
  Interventions: Device: MD Tissue Collagen Medical Device

INTERVENTIONS:
Device: MD Tissue Collagen Medical Device — The Experimental Group will be treated with 2-mL volume ultrasound-guided infiltration of: MD-Tissue (GUNA, Milan-Italy). Composition for 2 ml: collagen 100 micrograms Subjects will be treated with No.1 infiltration per week for 3 consecutive weeks. The infiltrations will be performed in an echoguided mode.
  MD-Tissue Collagen Medical Device will be infiltrated into the trochanteric bursa and at the level of the tendons of the gluteus minimus and gluteus medius, particularly at the level of the most degenerated insertional areas.

SUMMARY:
Greater Trochanteric Pain Syndrome, also known as GTPS (Greater Trochanteric Pain Syndrome) is a complex clinical condition characterized by chronic and recurrent pain in the lateral region of the hip, near the greater trochanter of the femur.

Biomechanical and anatomic-histologic interactions of the structures of the peri trochanteric space, in which, given the close anatomic-functional relationships, the origin can be traced to three different pathologic entities that may influence each other and fuel the progressive exacerbation of symptomatology. These are: external snap hip, trochanteric bursitis, and tendinopathies of the tendons of the gluteus mediums and gluteus minimums muscles.

Recent studies regarding GTPS have shown that in most cases this condition is due to degenerative tendinopathy of the tendons of the gluteus minimums and gluteus mediums muscles. Tendinopathy is defined as a pathological condition associated with histological changes that may result in a change in the organization of collagen fibrils, relative increase in the percentage of proteoglycans, glycosaminoglycans, and no collagenous components of the ECM accompanied by neo-vascularization and inflammatory state.

Tendinopathies thus result in painful symptomatology that very often also results in biomechanical functional deficit.

Clinically, GTPS presents as pain that is often debilitating and exacerbated by activities such as walking, climbing stairs, and lying on the affected side at night, associated with a progressive loss of stenia in hip abduction movements. On objective examination, a point of tenderness (trigger point) is noted at the level of the region of the greater trochanter, which may radiate to the lumbar area and along the lateral aspect of the thigh to the ipsilateral knee and a difficulty on strength versus resistance tests in hip abduction movements.

Although it is a very common syndrome, the treatment of painful grand trochanter syndrome, as well as that of tendinopathies in general, is still a major hurdle because the specific cellular pathogenetic and biomechanical etiopathogenetic mechanisms are still partly unknown and many treatments are empirical. Traditionally, the treatment of GTPS is initially conservative and includes rest, ice, NSAIDs and physiotherapy with stretching exercises of the fascia late. The use of corticosteroids, with systemic or local infiltrative intake, for the treatment of tendinopathies is highly controversial and, in any case, does not seem to have long-term efficacy.

MD-Tissue Collagen Medical Device is an injectable medical device based on porcine collagen type I; the collagen content is 100µg/2mL. Porcine collagen is like human collagen and highly compatible; it has very low risks of inducing adverse effects and is therefore used in several clinical settings.

DETAILED DESCRIPTION:
This is a pilot monocentric Clinical Investigation based on a One sample design.

In the ex vivo study, MD-Tissue Collagen Medical Device was used as a substrate for cell cultures of human gluteal tenocytes on culture plates. The results suggest how MD-Tissue can induce an anabolic phenotype in tenocytes by stimulating their proliferation and migration; it would also be able to promote the synthesis, maturation, and secretion of COL-I, thereby promoting tendon homeostasis and repair. Specifically, the modification of gene expression and proteins involved in collagen turnover pathways were analyzed by real-time PCR, Slot blot and SDS-zymography. Data from the study showed that tenocytes cultured with MD-Tissue compared with controls exhibited increased secretion and migration of COL-1 increased mRNA levels of the matrix metalloprotease inhibitor proteins MMP-1 and TIMP-1.

The tenocytes used for the cell cultures were gluteal tenocytes, derived from human gluteal tendon fragments (obtained from subjects without any tendon pathology who had undergone total hip replacement surgery); therefore, it is reasonable to think that the porcine type I collagen-based compound may be a viable treatment in GTPS.

The results of the preclinical study suggest how MD-Tissue Collagen Medical Device can induce an anabolic phenotype in tenocytes by stimulating tenocyte proliferation and COL-I synthesis, maturation, and secretion, thereby promoting tendon repair. As these effects have been evaluated ex vivo on tenocytes of gluteal muscle tendons, the purpose of this study is to evaluate its efficacy in local infiltrative treatment, in the pertechnetic region, of GTPS, in terms of resolution of pain symptoms and recovery of stenia in abduction.

Variables will be assessed at 6 different times; at baseline (day 0), after week 1, weeks 2, weeks 6, weeks 10 and after weeks 24.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 70 years;
* subjects with lateral palpatory pain that has appeared for at least 1 month;
* subjects with hip pain symptomatology assessed by Numerical rating scale (NRS) ≥ to 5;
* Subjects able to cooperate for the assessments in the Survey plan;
* subjects able to understand and sign informed consent.

Exclusion Criteria:

* subjects with true coxalgia (with positive FADDIR);
* subjects with ESHS (external snap hip syndrome);
* subjects already undergoing candidate hip replacement surgery;
* subjects with radiologic and clinical evidence of small and/or middle gluteal tendon detachment with indication for surgical repair;
* subjects with evidence of radiographically documented tendon calcifications;
* subjects with a degree of coxarthrosis of the hip that is a candidate for treatment according to the classification of Tonnis>1
* subjects who have taken fluoroquinolones within 30 days prior to enrollment
* subjects who have undergone treatment with hyaluronic acid or corticosteroids in the hip candidate for infiltrative treatment within 4 weeks before enrollment;
* subjects with local infections of the treatment candidate hip or systemic infections, osteomyelitis, or sepsis;
* subjects on chronic treatment with corticosteroids or immunosuppressants;
* subjects who are drug addicts, alcoholics, have psychiatric disorders, or have clinical conditions that may compromise the correct interpretation of PROMs or follow-up;
* subjects with coagulopathies, platelet aggregation disorders, or on treatment with oral anticoagulants or antiplatelets that cannot be discontinued during the study period;
* Pregnant and lactating subjects (female subjects of childbearing age should be tested for pregnancy before enrollment);
* subjects with allergy to porcine collagen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randelli RFMN Filippo Maria Nicola, Prof, Principal Investigator — Gaetano Pini CTO
Locations (1):
- Gaetano Pini CTO, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MD Tissue Collagen Medical Device
Started | 47
Completed | 42
Not Completed | 5
Not completed — 4 drop out and one withdrawn | 5

BASELINE CHARACTERISTICS:
Arm/Group | MD-Tissue Medical Device
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in NRS (Numerical Rating Scale) Pain Score From Baseline (Week 0) to Week 10
Description: Pain intensity was measured using the NRS (Numerical Rating Scale), a validated scale ranging from 0 (no pain) to 10 (worst possible pain).
  Participants were asked to indicate their pain level at baseline (Week 0) and at Week 10.
  A change of at least 3 points on the NRS is considered clinically significant. The primary outcome is the mean change in NRS score from baseline to Week 10.
Time Frame: weeks 10
Population: All variables will be subjected to the appropriate descriptive analyses after validation of the input data. Continuous variables: mean ± standard deviation or median and range, depending on the distribution; categorical variables: absolute and relative frequency tables.
Measure: Mean (95% Confidence Interval); unit: NRS Pain Score (range 0-10; higher score
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 47
NRS Pain Score (range 0-10; higher score | 4.7 [4.01 to 6.93]

2. Secondary Outcome: Mean NRS (Numerical Rating Scale) Pain Score at Week 6 and Week 24 Compared to Baseline (T0)
Description: Pain intensity was measured using the NRS (Numerical Rating Scale) at rest, ranging from 0 (no pain) to 10 (worst possible pain). Participants were asked to rate their pain at baseline (T0), week 6 (T6w/FU), and week 24 (T24w/FU). This outcome reports the mean NRS values at week 6 and 24. Higher scores indicate more intense pain.
Time Frame: weeks 6 and weeks 24
Population: All variables were subjected to the appropriate descriptive analyses after validation of the input data. Continuous variables were analyzed as mean ± standard deviation or median and range, depending on the distribution. Categorical variables were summarized as absolute and relative frequency tables.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 47
score on a scale
  NRS Week 6 | 4.5 [4.04 to 4.96]
  NRS Week 24 | 2.5 [2.03 to 2.97]

3. Secondary Outcome: Change in Modified Harris Hip Score (mHHS) From Baseline to Weeks 6, 10, and 24
Description: The Modified Harris Hip Score (mHHS) is a validated tool for assessing hip function and pain. It ranges from 0 (worst functional outcome and highest pain) to 100 (best function and least pain). Participants were evaluated at Weeks 6, 10, and 24 compared to baseline. The change in total score is used to assess clinical improvement.
  Unit of Measure:
  Score from 0 to 100; higher scores indicate better outcome
Time Frame: Weeks 6, 10, and 24
Measure: Mean (Standard Deviation); unit: Score from 0 to 100; higher scores indic
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 43
Score from 0 to 100; higher scores indic
  T0 (Baseline) | 57.09 (13.78)
  T6w | 71.22 (11.92)
  T10w | 72.53 (12.26)
  T24w | 73.19 (12.74)

4. Secondary Outcome: Change in Hip Abduction Strength From Baseline to Weeks 6, 10, and 24
Description: Hip abduction strength was assessed using a handheld dynamometer at Weeks 6, 10, and 24. The measurement was performed with the patient standing on the contralateral (healthy) limb, while abducting the hip affected by GTPS. For each assessment, three consecutive measurements were taken and averaged. Results were compared to baseline (Day 0) to evaluate functional improvement in muscular strength.
Time Frame: Weeks 6, 10, and 24
Population: All patients who completed dynamometric testing at all timepoints (T0, T6, T10, T24) were included in the per-protocol analysis.
Measure: Mean (Standard Deviation); unit: Force in kg measured by handheld dynamom
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 43
Force in kg measured by handheld dynamom
  Row Title Number Analyzed Mean SD T0 | 5.538 (2.8413)
  T6 | 6.045 (2.4797)
  T10w | 6.676 (3.0115)
  T24w | 6.851 (2.9481)
Statistical Analysis 1: Comparison: MD Tissue Collagen Medical Device; Hip abduction strength was analyzed using repeated measures ANOVA. The assumption of sphericity was tested and Bonferroni correction was applied for pairwise comparisons. A p-value < 0.001 was considered statistically significant; Test type: Other — Repeated measures ANOVA; p = 0.001, ANOVA

5. Secondary Outcome: MRI Evaluation of Inflammatory and Degenerative Signs in the Peritrochanteric Region at Week 24 Compared to Baseline
Description: MRI evaluation focused on inflammatory and degenerative signs in the peritrochanteric region (gluteus medius/minimus tendons) was conducted at Week 24 and compared to baseline (Week 0). Two independent radiologists assessed peri-tendinous fluid and intra-tendinous edema on STIR-weighted images. Improvement was defined as visible reduction in peritendinous edema. The analysis was qualitative and dichotomous (Improved vs. Unchanged).
Time Frame: Week 24 compared to baseline (Week 0)
Population: Patients who underwent MRI evaluation both at baseline and at Week 24 were included in the analysis (n=40).
Measure: Number; unit: Participants with MRI improvement
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 40
Participants with MRI improvement | 40
Statistical Analysis 1: Comparison: MD Tissue Collagen Medical Device; MRI improvement was assessed using paired evaluation of inflammatory signs (edema) at baseline and Week 24. McNemar exact test was used for within-subject categorical comparison; Test type: Other — McNemar Exact Test; p < 0.0001, McNemar — P-value derived from McNemar exact test comparing binary outcome (improved vs. unchanged). Statistical significance threshold set at p < 0.05; McNemar Exact Test

6. Secondary Outcome: Change in Analgesic Drug Consumption (Paracetamol and/or Celecoxib) From Baseline to Week 24
Description: Analgesic drug consumption (paracetamol and/or celecoxib) was recorded using a patient diary at time points T0 (baseline), T1w, T2w, T6w/FU, T10w/FU, and T24w/FU. Each patient logged the number of analgesic doses consumed per week. The total number of doses per timepoint was used to assess any significant change over time. The analysis aimed to evaluate whether the treatment reduced the need for pain medication, as an indirect marker of clinical efficacy.
  Unit of measure: Number of analgesic doses consumed per week.
Time Frame: Week 1, Week 2, Week 6, Week 10, and Week 24 compared to baseline (Week 0) Week 1, Week 2, Week 6, Week 10, and Week 24 compared to baseline (Week 0) Week 1, Week 2, Week 6, Week 10, and Week 24 compared to baseline (Week 0)
Population: All participants who returned complete analgesic diaries at each visit (Weeks 1, 2, 6, 10, and 24) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units of analgesics consumed (number of
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 43
Units of analgesics consumed (number of
  Week 1 | 1.6 (1.8)
  Week 2 | 0.8 (1.4)
  Week 6 | 0.5 (1.2)
  Week 10 | 0.3 (0.9)
  Week 24 | 0.7 (2.6)
Statistical Analysis 1: Comparison: MD Tissue Collagen Medical Device; Analgesic use (units/week) was analyzed over time using the Friedman test for repeated measures. No significant variation across follow-up visits was found; Test type: Other — Friedman Test Within-group; p = 0.992, Friedman Test Within-group

7. Secondary Outcome: Incidence of Adverse Events (AE, SAE, SUSAR) From Baseline to Week 24
Description: Adverse events (AEs), serious adverse events (SAEs), and suspected unexpected serious adverse reactions (SUSARs) were monitored at each study visit from baseline (Day 0) to Week 24. Data were collected via systematic interviews and clinical assessments. No adverse events of any type were reported during the study. AE definitions followed ICH-GCP and ClinicalTrials.gov guidance.
Time Frame: Day 0 to Week 24
Measure: Number; unit: participants
Arm/Group | MD Tissue Collagen Medical Device
Number analyzed (Participants) | 43
participants
  All-Cause Mortality | 0
  Serious Adverse Events | 0
  Other (Non-Serious) Adverse Events | 0

ADVERSE EVENTS:
Time Frame: The occurrence of Adverse Events will be assessed at each visit. T 0, T 1, T2, T6, T10 e T24 Weeks.
Description: The definitions of adverse event and serious adverse event used in this study were consistent with the ClinicalTrials.gov definitions. No adverse events, serious or non-serious, were observed during the study.
Groups:
- MD Tissue Collagen Medical Devic: MD Tissue Collagen Medical Device Show Description The Experimental Group will be treated with 2-mL volume ultrasound-guided infiltration of: MD-Tissue...
Arm/Group | MD Tissue Collagen Medical Devic
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

LIMITATIONS AND CAVEATS:
The limitations are constituted by the monocentric nature, the short follow-up and the absence of PROMs dedicated to hip tendon pathology. This last factor could induce a ceiling effect at the mHHS. Larger studies with longer follow-ups are desirable to try to find a final solution to this ubiquitous and disabling pathology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05486078/Prot_SAP_002.pdf